CLINICAL TRIAL: NCT03070938
Title: A Prospective, Observational Study of the Use of PuraPly™ Antimicrobial in the Management of Wounds
Brief Title: PuraPly™ Antimicrobial Wound Matrix and Wound Management
Acronym: PuraPlyAM
Status: Completed | Type: Observational
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Other Study IDs: PuraPly AM Case Series
Record Dates: First submitted 2016-12-07; First posted 2017-03-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Pressure Ulcer; Venous Ulcer; Diabetic Ulcer; Surgical Wound; Trauma Wound
Keywords: Chronic wounds; Acute Wounds; PHMB; Wound Management; Bioburden; Collagen
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PuraPly™ Antimicrobial Wound Matrix — PuraPly AM consists of a collagen sheet coated with polyhexamethylenbiguanide hydrochloride (PHMB) intended for the management of wounds. PuraPly AM is supplied dry in sheet form. The device is packaged in sterile, sealed single patches.
  Other Names: PuraPly AM

SUMMARY:
The PuraPly Antimicrobial Wound Matrix (PuraPly AM) case series is a prospective, observational study for patients who have received PuraPly AM which consists of a collagen sheet coated with polyhexamethylenbiguanide hydrochloride (PHMB) and is intended for the management of wounds; no experimental intervention is involved.

DETAILED DESCRIPTION:
The purpose of the case series is to assess the ability of PuraPly AM to meet wound specific treatment goals including management of bioburden, support of granulation tissue formation and support of wound closure. Patients will undergo clinical assessments and receive the standard of care as determined by the treating physician.

The case series is being undertaken to better understand PuraPly AM utilization and subsequent healing outcomes as well as to evaluate the effects of concomitant wound therapy on healing. Patient's participation may involve follow-up for up to 12 weeks following application of PuraPly AM.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 18 years of age
2. Participant has read, understood and signed and Institutional Review Board (IRB) approved Informed Consent Form (ICF).
3. Participant has at least 1 wound appropriate for receiving PuraPly AM, including

   * Partial and full-thickness wounds
   * Pressure ulcers
   * Venous ulcers
   * Diabetic ulcers
   * Chronic vascular ulcers
   * Tunneled/undermined wounds
   * Surgical wounds (donor sites/grafts, post-Mohs' surgery, post-laser surgery, podiatric, wound dehiscence) h. Trauma wounds (abrasions, lacerations, second-degree burns, skin tears) i. Draining wounds

Exclusion Criteria:

1. Participant has a known sensitivity to porcine materials
2. Participant has a third-degree burn
3. Participant has a known sensitivity to polyhexamethylenbiguanide hydrochloride (PHMB)
4. Participants receiving concurrent treatment with other topical antimicrobials or skin substitute products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are men and women at least 18 years old, with an eligible target wound that meets the Investigator's wound specific treatment goals that include the management of bioburden, support of granulation tissue formation and support of wound closure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Improvement in wound bed condition | 12 Weeks
  As measured from change in status from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gorenstein, MD, Principal Investigator — Winthrop University Hospital/ Winthrop Wound Healing Center
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided